CLINICAL TRIAL: NCT03066895
Title: Development and Testing of BabyGentleStick™ Vibrated Needle System for Heel Lance- Neonatal Pilot Study
Brief Title: BGS Neonatal Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actuated Medical, Inc. (Industry)
Collaborators: Milton S. Hershey Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: STUDY00006878
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pain From Heel Sticks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): BabyGentleStick
  Interventions: Device: BabyGentleStick
- Standard of Care (Active Comparator): HMC Standard Lancing Device
  Interventions: Device: Standard Lancing Device

INTERVENTIONS:
Device: BabyGentleStick — Experimental device.
  Arms: Experimental
Device: Standard Lancing Device — HMC standard of care.
  Arms: Standard of Care

SUMMARY:
This is a pilot, randomized, safety and efficacy study of an investigational device (i.e. BabyGentleStick™; BGS, Actuated Medical, Inc). The primary study objectives are to obtain subject feedback, assess device performance; and ascertain potential harm in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable late preterm/term neonates with a gestational age at birth of > 35 weeks gestation at birth
* Sex: male or female

Exclusion Criteria:

* Congenital anomalies or conditions at birth impacting central nervous system functioning and autonomic measurements
* Known risk for bleeding (i.e. Hemophilia, blood clotting or protein disorders)
* Prolonged labor or delayed birth with evidence of perinatal depression (e.g. Infant Apgar scores below 5)
* Identified maternal opiate dependency during pregnancy placing the infant at risk for opiate withdrawal, also known as neonatal abstinence syndrome (NAS)
* Critical illness in the mother preventing the ability to obtain informed consent from parents

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 8 days
  No device-attributable adverse events.

SECONDARY OUTCOMES:
Pain Response | 2 minute intervals, starting at 15 minutes before procedure and continuing until 10 minutes post procedure
  Pain level at specified study intervals measured on Neonatal Facial Coding System (NFCS) scale

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Clement, Ph.D., Principal Investigator — Actuated Medical, Inc.; Kim Doheny, Ph.D., Principal Investigator — The Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No